CLINICAL TRIAL: NCT07296237
Title: DACG VI. Beyond Survival: Addressing Gynecological and Sexual Health in Women After Radiotherapy for Anal Cancer
Brief Title: Beyond Survival: Addressing Gynecological and Sexual Health in Women After Radiotherapy for Anal Cancer
Acronym: DACG VI
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Department of Oncology, Vejle Hospital (Unknown); Department of Oncology Herlev Hospital, Denmark (Unknown)
Responsible Party: Principal Investigator, Johanne Hollands Steffensen, MD., Aarhus University Hospital
Other Study IDs: 1-10-72-19-25; 1-10-72-19-25 (Other: The Regional Ethics Committee for the Central Denmark Region)
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Anal Cancer
Keywords: anal cancer; Radiotherapy; Sexual dysfunction; Female sexual health; Gynecological side effects; Patient-reported outcomes
MeSH Terms: conditions — Anus Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
The goal of this observational study is to learn how radiotherapy for anal cancer affects the vaginal and sexual health of women after treatment. The study will also look at whether the radiation dose to the vagina is linked to the level of vaginal problems.

The main questions this study aims to answer are:

* How many women develop moderate or severe narrowing of the vagina after radiotherapy?
* Is there a link between the radiation dose and vaginal problems?
* How do vaginal changes affect sexual health and daily life?
* What care and support do women receive, and how satisfied are they with this support?

Participants are women aged 18 years or older who were treated with chemotherapy and radiotherapy for anal cancer and are 6 to 36 months after treatment.

Participants will:

Have a gynaecological examination to check the vagina for changes such as narrowing, stiffness, bleeding, or scarring Complete online questionnaires about quality of life and sexual health Answer questions about use of vaginal dilators, hormone treatment, and sexual counselling Allow researchers to analyse their radiotherapy scans to measure how much radiation the vagina received Some participants will also take part in a telephone interview about their experience with guidance and support after treatment

The study will include about 80 participants across three Danish hospitals. About 20 participants will take part in the interview part of the study.

The results from this study may help improve how doctors and nurses prevent, detect, and treat vaginal and sexual problems after radiotherapy for anal cancer. This may lead to better support and quality of life for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Diagnosed with anal cancer
* Treated with chemoradiotherapy with curative intent
* Between 6 and 36 months since completion of radiotherapy
* Able and willing to give written informed consent

Exclusion Criteria:

* Previous pelvic radiotherapy for another disease
* Treated with electron beam radiotherapy
* Unable to speak or understand Danish

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult women who have been treated with chemoradiotherapy for anal cancer in Denmark. Participants are recruited during routine follow-up visits at three oncology departments. All participants are between 6 and 36 months after treatment and are in cancer follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of moderate to severe vaginal stenosis after radiotherapy for anal cancer | Single assessment at study visit, 6 to 36 months after completion of chemoradiotherapy
  This outcome measures how many participants have moderate or severe narrowing of the vagina after treatment for anal cancer. Vaginal stenosis will be assessed during a gynaecological examination using a standard clinical grading system CTCAE v. 5.

SECONDARY OUTCOMES:
Gynecological findings at examination after radiotherapy for anal cancer | Single assessment at study visit, 6 to 36 months after completion of chemoradiotherapy
  This outcome measures physical changes in the vagina assessed during a standardised gynaecological examination. Findings include vaginal stiffness, scarring, fragile tissue with bleeding, small visible blood vessels, ulcers, and adhesions. All findings are recorded using a structured electronic clinical examination form based on established vaginal morbidity assessment methods.
Patient-reported sexual health and quality of life after radiotherapy for anal cance | Single assessment at study visit, 6 to 36 months after completion of chemoradiotherapy
  Participants complete validated questionnaires covering sexual health and quality of life:
  * EORTC QLQ-C30 and EORTC QLQ-ANL27 for general and anal cancer-specific quality of life
  * EORTC QLQ-SH22 for sexual health, including vaginal dryness, pain, and sexual satisfaction
  * Female Sexual Function Index (FSFI) for sexual desire, arousal, lubrication, orgasm, satisfaction, and pain
  All questionnaires use fixed response scales and are scored according to official scoring manuals.
Use of vaginal dilators, hormone treatment, and sexual counselling after radiotherapy | Single questionnaire assessment at study visit, 6 to 36 months after completion of chemoradiotherapy
  This outcome measures how often participants use vaginal dilators, whether they use local or systemic hormone treatment, and whether they have received specialised sexual counselling after radiotherapy. Data are collected using a structured pattern-of-care questionnaire completed by participants.
Radiation dose to the vagina and its relation to vaginal stenosis | Retrospective analysis of radiotherapy plans after study inclusion
  This outcome measures the radiation dose received by the vagina during treatment and examines its relation to moderate or severe vaginal stenosis. The vagina is outlined retrospectively on radiotherapy planning scans, and dose-volume data are extracted from treatment plans. These dose data are analysed in relation to clinical findings of vaginal stenosis.
Patient satisfaction with guidance on gynecological and sexual side effects | Single telephone interview within 3 months after study inclusion
  This outcome measures how satisfied participants are with the information and support they received about vaginal and sexual side effects after radiotherapy. Data are collected through semi-structured telephone interviews, which explore timing, clarity, and usefulness of the guidance. Interview data are analysed using thematic analysis.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Department of Oncology Aarhus University Hospital (AUH), Aarhus
  - Department of Oncology, Herlev and Gentofte Hospital, Herlev
  - Department of Oncology Vejle Hospital, University Hospital of Southern Denmark, Vejle

DOCUMENTS (1):
  • Study Protocol (2025-03-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT07296237/Prot_000.pdf